CLINICAL TRIAL: NCT02353442
Title: Biomechanical and Neurophysiological Changes in Subjects With Posterior Capsule Tightness - Evaluation and Treatment
Brief Title: Changes in Subjects With Posterior Capsule Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Dayana Patricia Rosa, Universidade Federal de São Carlos, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 860.648
Record Dates: First submitted 2015-01-18; First posted 2015-02-02 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Shoulder Pain
Keywords: Pain; Rotator cuff; Stretching; Mobilization; Scapula; Posterior capsule
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): This group will perform during 4 weeks:
  * placebo ultrasound during 5min ;
  * scapular squeezing in the sitting position (3x10repetitions);
  * upper trapezius stretching (in sitting position, 3x30s and 30s of rest).
  Interventions: Other: Placebo ultrasound; Other: Scapular squeezing; Other: Upper trapezius stretching
- Experimental group (Active Comparator): This group will perform during 4 weeks:
  * posterior shoulder mobilizations during 5min (mobilizations during 30s and 30s of rest);
  * external rotators strengthening in sidelying positions with load (3x10repetitions);
  * posterior capsule stretching (sleeper stretch in sidelying position, 3x30s and 30s of rest).
  Interventions: Other: Posterior shoulder mobilizations; Other: External rotators strengthening; Other: Posterior Capsule Stretching

INTERVENTIONS:
Other: Posterior shoulder mobilizations — A second investigator performed 5min of posterior capsule shoulder mobilization for the experimental group, 3times/week during 4 weeks.
  Arms: Experimental group
Other: External rotators strengthening — Individuals performed 3x10 repetitions of external rotators strengthening in sidelying position 3times/week during 4 weeks.
  Arms: Experimental group
Other: Placebo ultrasound — A second investigator performed 5min of placebo ultrassound for the control group, 3times/week during 4 weeks.
  Arms: Control group
Other: Scapular squeezing — Individuals performed 3x10 repetitions scapular squeezing exercise 3times/week during 4 weeks.
  Arms: Control group
Other: Upper trapezius stretching — Individuals performed 3x30s of upper trapezius stretching, 3times/week during 4 weeks.
  Arms: Control group
Other: Posterior Capsule Stretching — Individuals performed 3x30s of posterior capsule stretching, 3times/week during 4 weeks.
  Arms: Experimental group

SUMMARY:
To identify biomechanical and sensibility changes in people with posterior capsule tightness in people with and without shoulder pain.

DETAILED DESCRIPTION:
Some studies have shown that posterior capsule tightness can be related with shoulder dysfunctions and kinematics alterations. This study will be divided in two studies. The purpose of study 1 will be to assess the scapular and humeral kinematics, the strength of the shoulder external rotators and the pressure pain threshold in subjects with posterior capsule tightness with and without shoulder pain. Study 2 will verify the effects of two different treatments in subjects with posterior capsule tightness and shoulder pain on the same variables of study 1. One-hundred subjects will participate in the first study and will be divided in 4 groups: Group 1 - 25 subjects with shoulder pain and posterior capsule tightness; Group 2 - 25 subjects with no shoulder pain and no posterior capsule tightness; Group 3 - 25 subjects with shoulder pain and no posterior capsule tightness; and group 4 - 25 subjects with no shoulder pain and no posterior capsule tightness. All subjects will complete the DASH and Shoulder Pain and Disability Index questionnaires. External and internal rotation range of motion, strength of the external rotators, scapular kinematics and humeral translations during arm elevation, and pressure pain threshold will be measured. For the second study 50 subjects with shoulder pain and posterior capsule tightness will be recruited. The subjects will be randomly divided in 2 groups: experimental group or control group. The experimental group will receive glenohumeral posterior mobilization, stretching of posterior capsule and strengthening of the shoulder external rotators. The control group will do ultrasound;, stretching for the upper trapezius and scapular squeezing. Both groups will receive intervention for 3x/week/4 weeks. All subjects will be supervised for one physiotherapist and same variables from study 1 will be analyzed at pre and post-intervention.

ELIGIBILITY:
Inclusion Criteria: all subjects should have posterior capsule tightness and shoulder pain. So they should have:

* low flexion test (flexion + internal rotation) > 7°, between arms;
* symptoms consistent to shoulder impingement and arm elevation close to 150° as determined by digital inclinometer. The diagnosis for SIS was made based on a clinical examination and self-reported history. To be classified as having shoulder impingement, subjects had to present with at least 3 of the following: positive Neer test, positive Hawkins test, positive Jobe test, pain with passive or isometric resisted shoulder lateral rotation, pain with active shoulder elevation, and pain in the anterolateral shoulder region.

Exclusion Criteria: Individuals from both groups were excluded if they:

* were pregnant;
* had ligamentous laxity based on positive Sulcus test, Apprehension test or anterior drawer;
* had history of clavicle, scapula or humerus fracture;
* history of shoulder surgery or traumatic lesion; -had adhesive capsulitis or scoliosis; - had systemic illnesses;
* transpore tape allergy;
* body mass index > 28kg/m2;
* physical therapy treatment in the last 6 months;
* bilateral symptoms;
* steroid injection in the last 6 weeks;
* drugs with muscle relaxant in the last 72 hours.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dayana Rosa, Ms, Principal Investigator — UFSCar
Locations (1):
- UFSCar, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participation of all subjects was voluntary and no incentives were given to encourage enrollment. Fliers posted in the local university setting and surrounding community were used to recruit individuals from March 2015 to March 2016.
Groups:
- Control Group: This group will perform during 4 weeks:
  * placebo ultrasound during 5min ;
  * scapular squeezing in the sitting position (3x10repetitions);
  * upper trapezius stretching (in sitting position, 3x30s and 30s of rest).
  Posterior shoulder mobilizations: The subjects will be randomized to Experimental or control group.
- Experimental Group: This group will perform during 4 weeks:
  * posterior shoulder mobilizations during 5min (mobilizations during 30s and 30s of rest);
  * external rotators strengthening in sidelying positions with load (3x10repetitions);
  * posterior capsule stretching (sleeper stretch in sidelying position, 3x30s and 30s of rest).
  Posterior shoulder mobilizations: The subjects will be randomized to Experimental or control group.
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 28 | 31
Completed | 25 | 27
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 31 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.08 (12.08) | 41.18 (12.84) | 40.63 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 15 | 23 | 38
Region of Enrollment [Number; unit: participants]
  Brazil | 28 | 31 | 59

OUTCOME MEASURES:

1. Primary Outcome: Scapular Kinematics at 4weeks (Pre and Post Treatment)
Description: It was assessed in degrees with 3D system pre and post treatment.
Time Frame: 4 weeks: Baseline (pre-treatment), and 4 weeks (post-treatment)
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 27
degrees
  Pre Internal Rotation | 34.58 (0.69) | 36.00 (0.68)
  Post Internal Rotation | 34.76 (0.79) | 35.72 (0.77)
  Pre Upward Rotation | -18.12 (0.68) | -16.47 (0.66)
  Post Upward Rotation | -17.85 (0.58) | -14.37 (0.57)
  Pre Posterior Tilt | -3.23 (0.59) | -2.41 (0.58)
  Post Posterior Tilt | -3.66 (0.60) | -2.27 (0.59)

2. Primary Outcome: Humeral Translations at 4weeks (Pre and Post Treatment).
Description: It was assessed in millimeters with 3D system pre and post treatment.
Time Frame: 4 weeks: Baseline (pre-treatment), and 4 weeks (post-treatment)
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 27
Millimeters
  Pre Anterior Translation | 1.22 (0.36) | 0.85 (0.35)
  Post Anterior Translation | 0.68 (0.32) | 0.96 (0.32)
  Pre Superior Translation | 1.38 (0.28) | 1.21 (0.27)
  Post Superior Translation | 1.12 (0.22) | 0.66 (0.22)

3. Secondary Outcome: Strength of the Shoulder External Rotators at 4weeks (Pre and Post Treatment).
Description: The strength was evaluated with digital dynamometer in Newton pre and post treatment.
Time Frame: 4 weeks: Baseline (pre-treatment), and 4 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 27
Newton
  Pre External rotators strength | 89.08 (32.86) | 90.96 (28.71)
  Post External rotators strength | 88.98 (34.73) | 94.71 (27.59)

4. Secondary Outcome: Pressure Pain Threshold at 4weeks (Pre and Post Treatment).
Description: It was measured by a digital algometer in kPa pre and post treatment.
Time Frame: 4 weeks: Baseline (pre-treatment), and 4 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 27
kPa
  Pre Upper Trapezius | 287.40 (90.52) | 312.12 (135.02)
  Post Upper Trapezius | 351.47 (174.59) | 355.82 (161.77)
  Pre Infraspinatus | 351.33 (129.94) | 409.46 (198.58)
  Post Infraspinatus | 403.25 (211.70) | 438.51 (189.71)
  Pre Supraspinatus | 259.15 (86.68) | 321.07 (133.72)
  Post Supraspinatus | 343.88 (159.75) | 353.40 (161.16)
  Pre Deltoid | 301.78 (92.58) | 310.90 (147.84)
  Post Deltoid | 338.00 (149.94) | 344.56 (143.10)
  Pre Levator Scapulae | 256.63 (85.43) | 261.14 (125.89)
  Post Levator Scapulae | 267.26 (108.97) | 269.25 (109.36)
  Pre Anterior Tibialis | 711.31 (227.74) | 676.57 (270.60)
  Post Anterior Tibialis | 714.12 (272.46) | 748.09 (256.98)

5. Secondary Outcome: Pain and Function at 4weeks (Pre and Post Treatment)
Description: For these measures, the SPADI (Shoulder Pain and Disabilities Index) questionnaire was used, pre and post treatment. The is a self-assessment questionnaire with 5 questions about pain and 8 about functional activities. The final score (0-100) of the questionnaire is provided in percentage and a maximum score of 100 implies the worst possible condition.
Time Frame: 4 weeks: Baseline (pre-treatment), and 4 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 25 | 27
scores on a scale
  Pre SPADI score | 46.01 (24.11) | 45.26 (23.22)
  Post SPADI score | 27.10 (23.75) | 17.22 (15.04)

ADVERSE EVENTS:
Time Frame: 2 days after the pre and post evaluations.
Description: The Adverse Events were assessed, but they were not observed in this study
Arm/Group | Control Group | Experimental Group
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 0/28 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes